CLINICAL TRIAL: NCT04442113
Title: Multicenter Randomized Controlled Trial Assessing Targeted Ablation in Persistent Atrial Fibrillation Using the Stochastic Trajectory Analysis of Ranked Signals (STAR Mapping™) Method.
Brief Title: RandOmised Controlled Trial of STAR Mapping™ Guided Ablation for AF.
Acronym: ROC-STAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study cancelled. Different direction pursued by Rhythm AI.
Sponsor: Rhythm AI Ltd (Industry)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROC-STAR
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Catheter ablation; Arrhythmia; Cardiac mapping
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Pulmonary vein isolation alone (by catheter ablation)
  Interventions: Procedure: Pulmonary vein isolation
- STAR guided ablation group (Experimental): Pulmonary vein isolation plus ablation guided by STAR MappingTM
  Interventions: Procedure: Pulmonary vein isolation plus ablation guided by novel STAR mapping™

INTERVENTIONS:
Procedure: Pulmonary vein isolation plus ablation guided by novel STAR mapping™ — Catheter ablation for persistent AF consisting of pulmonary vein isolation plus additional ablation guided by the novel STAR mapping™ software on a computer device.
  Arms: STAR guided ablation group
Procedure: Pulmonary vein isolation — Catheter ablation for persistent AF consisting of pulmonary vein isolation (the standard treatment for AF)
  Arms: Control group

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia with an expected rise in prevalence over the next decade. Beyond causing troublesome symptoms AF is associated with increased mortality and morbidity. Catheter ablation is a safe treatment which is effective for paroxysmal AF but the success rate for persistent AF remains approximately 50% at 1 year. A new mapping technique, called Stochastic Trajectory Analysis of Ranked signals (STAR Mapping™) Method, has recently been developed. In a pilot study, localised sources driving AF were consistently mapped and ablated with excellent acute and long term outcomes. This trial will test the clinical effectiveness of this approach by comparing conventional ablation with pulmonary vein isolation (PVI) to PVI plus STAR mapping™ guided ablation. We plan to test this through a prospective multicenter randomized controlled trial including 177 patients.

DETAILED DESCRIPTION:
This will be a prospective multi-centre randomised controlled trial with two treatment arms. We plan to include up to 15 UK centres. Patients that have been referred for catheter ablation of symptomatic persistent AF will be recruited. Patients will be consented and have their baseline review after having been listed for AF ablation on the hospital waiting list. They will be randomized to one of two treatment arms. All patients will undergo their procedure using a 3D mapping system. Standard catheters will be used during the ablation procedure. Because the STAR mapping™ system will be configured for use with a special version of the 3D mapping system Carto (BIosense Webster) the study will mandate use of clinically approved Carto catheters: Smarttouch thermocool ablation catheter and the Pentarray mapping catheter. Ablation procedures will be carried out using the usual policies and protocols of the institutions involved except for the specific points below. The two treatment arms include:

1. Control arm - PVI alone After PVI, no further ablation in AF will be allowed. If the patient organizes into an atrial tachycardia (AT) during PVI this will be mapped and ablated. Otherwise, in accordance with common clinical practice, a 30 minute waiting period will be observed following PVI to watch for acute pulmonary vein reconnection. During this waiting period, mapping data will be acquired using the multipolar pulmonary vein mapping catheter to acquire STAR mapping™ data. The operator will be blinded to these data. This is done using the pentarray mapping catheter to acquire a minimum of 10 widely spaced globally distributed left atrial recordings of 30 seconds each outside the pulmonary veins. If the patient has remained in AF post PVI then electrical cardioversion will be performed, the pulmonary veins checked and re-isolated if needed, and the procedure terminated.
2. Experimental arm - PVI followed by STAR guided ablation. If the patient organises to sinus rhythm after PVI alone then a 30 minute wait will be observed to ensure sustained PVI and the procedure terminated. If patients remain in AF following PVI, the left atrium will be mapped using a multipolar mapping catheter to acquire a minimum of 10 widely spaced globally distributed recordings outside the pulmonary veins. STAR mapping™ data will be exported and maps generated. Ablation will then be targeted at the leading sites identified by STAR mapping™ in order of ranking (1st first, 2nd second, etc.) with the end-point of AF termination. If AF terminates further sites will not be targeted. If patients terminate to an atrial tachycardia then this will be mapped and ablated as per standard clinical practice.

If AF persists following ablation of all STAR mapping™ identified sites then mapping of the right atrium may be considered if the septum consistently activates early and the coronary sinus activation is predominantly proximal to distal, and further ablation permitted in the right atrium if indicated. If patients remain in AF following ablation then they will be electrically cardioverted.

Follow-up All patients will undergo 12 months follow-up with an ECG at 3, 6, 9 and 12 months, and a 48h ambulatory Holter monitor at 6 and 12 months. Patients will routinely continue anti-arrhythmic therapy for up to 3 months post procedure which will be considered a blanking period. After 3 months rhythmically active antiarrhythmic drugs will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* Persistent AF (continuous AF duration between 1 week and 24 months)
* No previous AF ablation or other left atrial ablation
* Undergoing a clinical AF ablation procedure.

Exclusion Criteria:

* Unwillingness to sign consent
* Any other contraindication to catheter ablation
* Age <18 years or > 80 years
* AF with a reversible cause
* AF that is paroxysmal
* AF that has been persistent > 2 yrs
* Previous left atrial ablation (percutaneous or surgical)
* Severe LV impairment (EF < 40%)
* NYHA class 3 or 4 heart failure
* Severely dilated left atrium (LA diameter > 50 mm)
* Known cardiomyopathy or inherited 'channelopathy'
* Congential heart disease (excluding PFO)
* More than moderate valvular heart disease or prosthetic heart valves
* Prior MI, PCI or cardiac surgery in the last 6 months
* Pregnancy
* Morbid obesity (defined as BMI >40)
* Any other medical problem likely to cause death within the next 18 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of subjects in the 2 groups with clinical success | 12 months
  Clinical success is defined as freedom from atrial arrhythmia (AF or atrial tachycardia) lasting >30 seconds after a single procedure off antiarrhythmic drugs subsequent to a 3 month blanking period (standard guideline definition of clinical success).
Comparison of the proportion of subjects in the 2 groups with termination of AF during ablation | During the index procedure (i.e. day 0)
  Termination of AF during ablation

SECONDARY OUTCOMES:
Comparison of the proportion of subjects in the 2 groups with major complications following their index procedure. | 30 days
  major complications are defined as any complication causing death, disability, results in another intervention, or prolongs hospital stay (as per guidelines).
Comparison of the proportion of subjects in the 2 groups with early failure following their index procedure. | 3 months
  Early failure is described as recurrent AF or atrial tachycardia at the 3 months time point.
Comparison of the proportion of subjects in the 2 groups reaching a composite electrophysiological end point during their index procedure | During the index ablation procedure (i.e. day 0)
  The composite electrophysiological end point is comprised of either AF termination or slowing of AF cycle length ≥30ms measured from the left atrial appendage during ablation.
Radiofrequency ablation time | Intraprocedural
  Duration of radiofrequency ablation
Procedure time | Intraprocedural
  Duration of procedure
Comparison of the proportion of subjects in the 2 groups with freedom from AF | 12 months
  Freedom from AF defined as no documented AF (>30 seconds) following the 3 months blanking period following a single procedure, off anti-arrhythmic drugs.
Comparison of the proportion of subjects in the 2 groups with freedom from atrial arrhythmia allowing for antiarrhythmic drugs. | 12 months
  Freedom from documented atrial arrhythmia (>30 seconds) following the 3 months blanking period following a single procedure, allowing for anti-arrhythmic drugs.
Comparison of the proportion of subjects in the 2 groups with freedom from AF allowing for antiarrhythmic drugs | 12 months
  Freedom from AF defined as no documented AF (>30 seconds) following the 3 months blanking period following a single procedure, allowing for anti-arrhythmic drugs.
Relationship between the number of AF drivers identified using STAR mapping™ and clinical outcome | 12 months
  The number of AF drivers identified will be correlated to the proportion of patients with clinical success at 1 year (the primary end-point). This analysis will be performed for all 177 patients, and for each of the 2 groups separately.

REFERENCES:
- [Background] Honarbakhsh S, Hunter RJ, Finlay M, Ullah W, Keating E, Tinker A, Schilling RJ. Development, in vitro validation and human application of a novel method to identify arrhythmia mechanisms: The stochastic trajectory analysis of ranked signals mapping method. J Cardiovasc Electrophysiol. 2019 May;30(5):691-701. doi: 10.1111/jce.13882. Epub 2019 Mar 5. PMID 30801836
- [Background] Honarbakhsh S, Hunter RJ, Ullah W, Keating E, Finlay M, Schilling RJ. Ablation in Persistent Atrial Fibrillation Using Stochastic Trajectory Analysis of Ranked Signals (STAR) Mapping Method. JACC Clin Electrophysiol. 2019 Jul;5(7):817-829. doi: 10.1016/j.jacep.2019.04.007. Epub 2019 May 8. PMID 31320010
- [Background] Honarbakhsh S, Schilling RJ, Finlay M, Keating E, Ullah W, Hunter RJ. STAR mapping method to identify driving sites in persistent atrial fibrillation: Application through sequential mapping. J Cardiovasc Electrophysiol. 2019 Dec;30(12):2694-2703. doi: 10.1111/jce.14201. Epub 2019 Oct 3. PMID 31552697
- [Background] Honarbakhsh S, Schilling RJ, Keating E, Finlay M, Hunter RJ. Drivers in AF colocate to sites of electrogram organization and rapidity: Potential synergy between spectral analysis and STAR mapping approaches in prioritizing drivers for ablation. J Cardiovasc Electrophysiol. 2020 Jun;31(6):1340-1349. doi: 10.1111/jce.14456. Epub 2020 Apr 9. PMID 32219906
- See also: Rhythm AI Ltd website — https://rhythm-ai.com/